CLINICAL TRIAL: NCT03799159
Title: Renal Arterial Resistive Index Versus Novel Serum and Urinary Biomarkers for Early Prediction of Sepsis Associated-acute Kidney Injury in Critically Ill Patients
Brief Title: Renal Arterial Resistive Index Versus Novel Biomarkers for Early Prediction of Sepsis Associated-acute Kidney Injury
Acronym: RRIBIOSAKI
Status: Completed | Type: Observational
Sponsor: Islam Elsayed Mohamed Ahmed (Other)
Responsible Party: Sponsor-Investigator, Islam Elsayed Mohamed Ahmed, Critical Care Clinical Pharmacy Specialist, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: RRIBIOSAKI
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Sepsis; Septic Shock; Acute Kidney Injury
Keywords: Sepsis; Acute Kidney Injury; Ultrasound; Resistive Index; Biomarkers
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for neutrophil gelatinase-associated lipocalin (NGAL) and Cystatin C (CysC).
  Urine samples for neutrophil gelatinase-associated lipocalin (NGAL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Populations at high risk of Sepsis-Associated Acute Kidney Injury (SA-AKI) have been identified. Sources of sepsis, in particular, bloodstream infection, abdominal and genitourinary sepsis, and infective endocarditis, are associated with a higher likelihood of developing AKI. Similar to the poor outcome of patients with sepsis, delayed administration of appropriate antimicrobial therapy was shown to be an independent predictor of the development of AKI. Incremental delays in antimicrobial delivery after the onset of hypotension showed a direct relationship with the development of AKI. The need for sensitive, simple and time-applicable biomarker to predict AKI development after renal insult is urgent.

Serum creatinine (sCr) and urea are used routinely for the diagnosis of AKI. However, these parameters are not accurate for the diagnosis of AKI. Cystatin C. (CysC) is suggested to be a good biomarker because of its constant rate of production, almost filtered by glomeruli (99%), has no significant protein binding and not secreted by renal tubule. Neutrophil gelatinase-associated lipocalin (NGAL) is recently identified and extensively investigated as a most promising early marker of AKI. Urinary NGAL is not only effective in detection of AKI but also its degree of expression might distinguish among AKI, prerenal azotemia and chronic kidney disease, and it is detectable before the accumulation of serum creatinine.

Ultrasonography (US) is used routinely to assess renal morphology. Renal Resistive Index (RRI) is a non-invasive Doppler-measured parameter that is directly correlated with intra-renal arterial resistance. RRI is defined as [(peak systolic velocity - end diastolic velocity)/ peak systolic velocity]. It theoretically ranges from 0 to 1 and it is normally lower than 0.7 with age differences. RRI calculation was found to be useful as an early indicator of the vascular resistance changes and in the determination of the optimal systemic hemodynamics required for renal perfusion.

The aim of this study is to compare the ability of arterial renal resistive index (RRI), serum and urinary neutrophil gelatinase-associated lipocalin (NGAL), Cystatin C (CysC) in early diagnosis and predicting the persistence of acute kidney injury in septic patients.

DETAILED DESCRIPTION:
All included patients in this study will be assessed for the following:

1. Data Collection

   * Complete history taking (age, sex, illness, medications, etc.).
   * Complete physical examination (Glasgow coma scale (GCS), temperature, blood pressure, urine output, heart rate, respiratory rate and chest auscultation).
   * SOFA score, APACHE II score, and Quick SOFA (qSOFA).
   * Routine laboratory investigations and Coagulation profile.
   * C-reactive protein (CRP), and Serum lactate.
   * Complete sepsis workup (chest x-ray, urine analysis, abdomen and pelvis ultrasound, microbiological cultures) to identify the source of sepsis.
2. Renal Biomarkers

   - Serum and urinary samples will be collected directly at time of enrollment (within 2 hours from admission). It will be assayed for serum creatinine, serum neutrophil gelatinase-associated lipocalin (NGAL), urinary NGAL and serum Cystatin C (CysC). Then, it will be repeated at day 3.
3. Ultrasound evaluation of kidneys and renal Doppler

   * In each patient, both kidneys will be examined with real-time ultrasound (US) with a 3.75-MHz transducer (ACUSON X 300). Pulsed Doppler US evaluation of the intrarenal arteries will be obtained at the same respective scanning frequencies. The color Doppler functions are set for a study focused on interlobar arteries, that is, the highest gains possible, the use of the lowest filters and a low pulse repetition frequency (PRF) of 1-1.5 kHz that must be preferred while always limiting the aliasing phenomenon.
   * The renal resistance index (RRI, [peak systolic frequency shift-minimum diastolic frequency shift]/ peak systolic frequency shift) will be calculated from calibrated software. (26) All measurements will be performed by the same examiner.
   * The renal resistive index (RRI) will be measured at time of enrollment (within 2 hours from admission) and 24 hours after admission.
4. Treatment All patients will receive the standard treatment for management of sepsis on the guidelines of SCC (sepsis-3). The protocol of treatment will not be changed during the study time.
5. Follow up - All patients will be followed up using urine output (UOP), serum creatinine, KDIGO (Kidney Disease Improving Global Outcomes) classification, the use of vasopressors and need for renal replacement therapy (RRT).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged above 18 years) recently admitted with sepsis

Exclusion Criteria:

* Pregnant Females
* Patients with renal transplant.
* Patients with End Stage Renal Disease (ESRD).
* Patients with Chronic Kidney Disease (CKD) known with history, laboratory or ultrasonographic evaluation with chronic nephropathic changes.
* Patients with renal artery stenosis.
* Patients with obstructive uropathy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Critically ill patients recently admitted with sepsis.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | 7 days from inclusion
  AKI is defined according to KDIGO (Kidney Disease Improving Global Outcomes)
Transient Acute Kidney Injury | 7 days from inclusion
  Transient AKI is defined as AKI with a cause of renal hypoperfusion and recovery within 3 days after inclusion. Recovery from AKI is defined as urine output normalization and/or serum creatinine decrease by 50% and/or serum creatinine normalization to its measured or estimated baseline level.
Persistent Acute Kidney Injury | 7 days from inclusion
  Persistent AKI is defined as persistent serum creatinine rise or oliguria after 3 days.

SECONDARY OUTCOMES:
Mortality | 28 days from inclusion
  All cause 28-days mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Ibrahim, MSc, Principal Investigator — Assistant Lecturer of Critical Care Medicine, Kafr Elsheikh University; Taysser Zaitoun, MD, Study Director — Professor of Critical Care Medicine, Alexandria University; Mohamed Megahed, MD, Study Director — Professor of Critical Care Medicine, Alexandria University; Hisham Elghonemy, MD, Study Chair — Lecturer of Nephrology, Alexandria University; Doaa Emara, MD, Study Chair — Lecturer of Radiodiagnosis, Alexandria University; Islam Ahmed, PharmD, Study Chair — Clinical Pharmacy Specialist, Alexandria University
Locations (1):
- Alexandria Main University Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
The summary of all relevant data

REFERENCES:
- [Background] Bagshaw SM, George C, Bellomo R; ANZICS Database Management Committee. Early acute kidney injury and sepsis: a multicentre evaluation. Crit Care. 2008;12(2):R47. doi: 10.1186/cc6863. Epub 2008 Apr 10. PMID 18402655
- [Background] Bagshaw SM, Uchino S, Bellomo R, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Oudemans-van Straaten HM, Ronco C, Kellum JA; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Septic acute kidney injury in critically ill patients: clinical characteristics and outcomes. Clin J Am Soc Nephrol. 2007 May;2(3):431-9. doi: 10.2215/CJN.03681106. Epub 2007 Mar 21. PMID 17699448
- [Background] Bagshaw SM, Lapinsky S, Dial S, Arabi Y, Dodek P, Wood G, Ellis P, Guzman J, Marshall J, Parrillo JE, Skrobik Y, Kumar A; Cooperative Antimicrobial Therapy of Septic Shock (CATSS) Database Research Group. Acute kidney injury in septic shock: clinical outcomes and impact of duration of hypotension prior to initiation of antimicrobial therapy. Intensive Care Med. 2009 May;35(5):871-81. doi: 10.1007/s00134-008-1367-2. Epub 2008 Dec 9. PMID 19066848
- [Background] Schnell D, Deruddre S, Harrois A, Pottecher J, Cosson C, Adoui N, Benhamou D, Vicaut E, Azoulay E, Duranteau J. Renal resistive index better predicts the occurrence of acute kidney injury than cystatin C. Shock. 2012 Dec;38(6):592-7. doi: 10.1097/SHK.0b013e318271a39c. PMID 23042202
- [Background] Merrikhi A, Gheissari A, Mousazadeh H. Urine and serum neutrophil gelatinase-associated lipocalin cut-off point for the prediction of acute kidney injury. Adv Biomed Res. 2014 Jan 27;3:66. doi: 10.4103/2277-9175.125847. eCollection 2014. PMID 24627874
- [Background] Zhang Z, Lu B, Sheng X, Jin N. Cystatin C in prediction of acute kidney injury: a systemic review and meta-analysis. Am J Kidney Dis. 2011 Sep;58(3):356-65. doi: 10.1053/j.ajkd.2011.02.389. Epub 2011 May 20. PMID 21601330
- [Background] Mori K, Lee HT, Rapoport D, Drexler IR, Foster K, Yang J, Schmidt-Ott KM, Chen X, Li JY, Weiss S, Mishra J, Cheema FH, Markowitz G, Suganami T, Sawai K, Mukoyama M, Kunis C, D'Agati V, Devarajan P, Barasch J. Endocytic delivery of lipocalin-siderophore-iron complex rescues the kidney from ischemia-reperfusion injury. J Clin Invest. 2005 Mar;115(3):610-21. doi: 10.1172/JCI23056. PMID 15711640
- [Background] Mishra J, Dent C, Tarabishi R, Mitsnefes MM, Ma Q, Kelly C, Ruff SM, Zahedi K, Shao M, Bean J, Mori K, Barasch J, Devarajan P. Neutrophil gelatinase-associated lipocalin (NGAL) as a biomarker for acute renal injury after cardiac surgery. Lancet. 2005 Apr 2-8;365(9466):1231-8. doi: 10.1016/S0140-6736(05)74811-X. PMID 15811456
- [Background] Nickolas TL, O'Rourke MJ, Yang J, Sise ME, Canetta PA, Barasch N, Buchen C, Khan F, Mori K, Giglio J, Devarajan P, Barasch J. Sensitivity and specificity of a single emergency department measurement of urinary neutrophil gelatinase-associated lipocalin for diagnosing acute kidney injury. Ann Intern Med. 2008 Jun 3;148(11):810-9. doi: 10.7326/0003-4819-148-11-200806030-00003. PMID 18519927
- [Background] Zwiers AJ, de Wildt SN, van Rosmalen J, de Rijke YB, Buijs EA, Tibboel D, Cransberg K. Urinary neutrophil gelatinase-associated lipocalin identifies critically ill young children with acute kidney injury following intensive care admission: a prospective cohort study. Crit Care. 2015 Apr 21;19(1):181. doi: 10.1186/s13054-015-0910-0. PMID 25895828
- [Background] Haase-Fielitz A, Bellomo R, Devarajan P, Bennett M, Story D, Matalanis G, Frei U, Dragun D, Haase M. The predictive performance of plasma neutrophil gelatinase-associated lipocalin (NGAL) increases with grade of acute kidney injury. Nephrol Dial Transplant. 2009 Nov;24(11):3349-54. doi: 10.1093/ndt/gfp234. Epub 2009 May 27. PMID 19474273
- [Background] Schnell D, Darmon M. Renal Doppler to assess renal perfusion in the critically ill: a reappraisal. Intensive Care Med. 2012 Nov;38(11):1751-60. doi: 10.1007/s00134-012-2692-z. Epub 2012 Sep 22. PMID 23001447
- [Background] Bougle A, Duranteau J. Pathophysiology of sepsis-induced acute kidney injury: the role of global renal blood flow and renal vascular resistance. Contrib Nephrol. 2011;174:89-97. doi: 10.1159/000329243. Epub 2011 Sep 9. PMID 21921613